CLINICAL TRIAL: NCT00227890
Title: Motivation and Skills for THC/ETOH+ Teens in Jail
Brief Title: Skills and Motivation at the Rhode Island Training School (Project SMART) - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lynda Stein, Ph.D., Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18851-1; R01DA018851 (NIH); R01-18851-1
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Alcoholic, Marijuana Misuse
Keywords: substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Motivational Interviewing followed by Cognitive Behavior Therapy (MI/CBT)
  Interventions: Behavioral: MI/CBT
- 2 (Experimental): Relaxation Training followed by Treatment as Usual (RT/TU)
  Interventions: Behavioral: RT/TU

INTERVENTIONS:
Behavioral: MI/CBT
  Arms: 1
Behavioral: RT/TU
  Arms: 2

SUMMARY:
This study will focus on treating substance abusing incarcerated teens using individually administered Motivational Interviewing (MI) followed by group Cognitive Behavior Therapy (CBT). The control group receives individualized Relaxation Training (RT) followed by group Treatment as Usual (TU). Currently, there is little research regarding effective group treatments for incarcerated teens and this study will address this gap in our knowledge base. We seek to reduce substance use and associated risky behaviors post-release (including driving under the influence, risky sexual behaviors, etc.).

DETAILED DESCRIPTION:
This proposal is in response to RFA-DA-04-008, Group Treatment for Individuals in Drug Abuse or Alcoholism Treatment. Of particular interest to the agencies are group therapies for Conduct Disordered adolescents, reducing the spread of infectious disease, and mechanisms of action. This proposal targets these areas of interest. This study will focus on treating substance abusing incarcerated teens using 2 individually administered Motivational Interviewing (MI) sessions followed by 10 group sessions of Cognitive Behavior Therapy (CBT). MI is conceptualized as preparation for group CBT. The control group receives individualized Relaxation Training (RT) followed by group Treatment as Usual (TU). Currently, there is little research regarding effective group treatments for incarcerated teens and this study will address this gap in our knowledge base.

In this proposed randomized trial, a one-way design (MI/CBT vs. RT/TU) will be used to determine whether MI/CBT enhances group therapy participation and reduces substance use and related problems (such as crime, injuries and unprotected sex) post discharge in substance-involved juvenile delinquents. RT/TU is based on the 12-step model and includes psycho-educational components. Participants are followed during incarceration and for 6 months post incarceration. Primary outcome variables include alcohol and marijuana use, as well as related behaviors (illegal activity, sex or injuries while drunk or high). It is hypothesized that in comparison to teens in RT/TU, youth receiving MI/CBT will participate more in therapy (according to teen, facility staff, and counselor ratings) and will show lower levels of substance use and related problems after discharge.

Frequently, substance abuse treatment is unavailable to youths in the juvenile justice system, and when treatment is available, it may be provided in group format using untested therapies. A motivation/skills-based intervention (delivered in group format) may prove efficacious in enhancing motivation and in reducing substance abuse and related problems. This study extends previous research by rigorously evaluating group treatment for incarcerated teens. We will examine processes contributing to the efficacy of group MI/CBT, and the influence of race and ethnicity on treatment effects. The development of effective interventions for substance using juvenile offenders has the potential to reduce substance abuse and crime in this population.

ELIGIBILITY:
Inclusion Criteria:

Adolescents will be eligible if in the year prior to incarceration they either a) drank alcohol or used marijuana at least once per month or b) binge-drank (> 5 for boys, < 4 for girls) during any two week period; or they drank or used marijuana in the four weeks before the offense for which they were incarcerated; or they used alcohol or marijuana in the four weeks before they were incarcerated.

Exclusion Criteria:

Those teens sentenced for less than 4 months or greater than 12 months, those who are younger than 14 years or older than 19 years, and those for whom have inability to consent/assent (example, language barrier) are not obtained will be excluded from participation.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 205 (Actual)
Dates: Start 2005-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Alcohol use, using Time-Line Followback, aggregated into quantity and frequency | 6 months post release
Marijuana use, using Time-Line Followback, aggregated into quantity and frequency | 6 months post release
Crime, using Misbehaviors Questionnaire, aggregated into type and frequency | 6 months post release

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Stein, Ph.D., Principal Investigator — University of Rhode Island
Locations (2):
- United States (2):
  - Rhode Island Training School, Cranston, Rhode Island
  - University of Rhode Island, Social Sciences Research Center, Kingston, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
With appropriate request and procedure.

REFERENCES:
- [Background] Stein LA, Clair M, Martin RA, Soenksen S, Lebeau R, Rohsenow DJ, Kahler CW, Hurlbut W, Monti PM. Measuring behaviors of individual adolescents during group-based substance abuse intervention. Subst Abus. 2014;35(4):408-17. doi: 10.1080/08897077.2014.949337. PMID 25127289
- [Background] Bernstein MH, Stein LA. Do bisexual girls report higher rates of substance use than heterosexual girls? A failure to replicate with incarcerated and detained youth. J Bisex. 2015;15(4):498-508. doi: 10.1080/15299716.2015.1057889. Epub 2015 Nov 17. PMID 27087787
- [Background] Martin RA, Stein LA, Clair M, Cancilliere MK, Hurlbut W, Rohsenow DJ. Adolescent Substance Treatment Engagement Questionnaire for Incarcerated Teens. J Subst Abuse Treat. 2015 Oct;57:49-56. doi: 10.1016/j.jsat.2015.04.011. Epub 2015 May 7. PMID 26021405
- [Background] Stein LA, Clair M, Rossi JS, Martin RA, Cancilliere MK, Clarke JG. Gender, ethnicity and race in incarcerated and detained youth: services and policy implications for girls. Psychiatr Rehabil J. 2015 Mar;38(1):65-73. doi: 10.1037/prj0000089. Epub 2014 Sep 1. PMID 25180525
- [Background] Stein LA, Clair M, Soenksen S, Martin RA, Clarke JG. Studying Process and Proximal Outcomes of Supervision for Motivational Interviewing. Train Educ Prof Psychol. 2015 May;9(2):175-182. doi: 10.1037/tep0000073. No abstract available. PMID 26417395
- [Background] Bassett SS, Stein LA, Rossi JS, Martin RA. Evaluating Measures of Fidelity for Substance Abuse Group Treatment With Incarcerated Adolescents. J Subst Abuse Treat. 2016 Jul;66:9-15. doi: 10.1016/j.jsat.2016.02.011. Epub 2016 Mar 9. PMID 27211991